CLINICAL TRIAL: NCT04762966
Title: Study of Metformin Overdose in Adult Patients Treated at the University Hospital of Nancy: Single-center Descriptive Retrospective Observational Study
Brief Title: Study of Metformin Overdose
Acronym: METINFO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, SCALA-BERTOLA Julien, Dr Julien SCALA-BERTOLA, Central Hospital, Nancy, France
Other Study IDs: 2021PI020
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Metformin Associated Lactic Acidosis
Keywords: Metformin; Lactic Acidosis; Causality assessment
MeSH Terms: conditions — Acidosis, Lactic | interventions — Metformin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Therapeutic: Patients with metformin blood concentration in the therapeutic ranges.
  Interventions: Drug: Metformin
- Supratherapeutic: Patients with metformin blood concentration above the therapeutic ranges.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Level of Metformin blood concentration

SUMMARY:
The objective of the METINFO study is an observational single-center retrospective and descriptive study. The main objective is to estimate the real mortality rate associated to a Metformin overdose. Second objectives are to estimate the real hospitalization rate related to metformin overdose and to identify the risk factors of a metformin overdose and especially the potential correlation between metformin blood concentration and overdose severity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients benifiting of a metformin blood concentration determination in the period ranging from the 1st of July 2019 and the 1st of July 2021.

Exclusion Criteria: None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients benifiting of a metformin blood concentration determination in the period ranging from the 1st of July 2019 and the 1st of July 2021 and hospitalized in the university hospital of Nancy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Estimation of Mortality Rate | 2 years

SECONDARY OUTCOMES:
Estimation of Hospitalization Rate | 2 years
Identification of Risk Factors | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nancy, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Background] Goonoo MS, Morris R, Raithatha A, Creagh F. Metformin-associated lactic acidosis: reinforcing learning points. BMJ Case Rep. 2020 Sep 2;13(9):e235608. doi: 10.1136/bcr-2020-235608. PMID 32878828
- [Background] Walz L, Jonsson AK, Ahlner J, Ostgren CJ, Druid H. Metformin - Postmortem fatal and non-fatal reference concentrations in femoral blood and risk factors associated with fatal intoxications. Forensic Sci Int. 2019 Oct;303:109935. doi: 10.1016/j.forsciint.2019.109935. Epub 2019 Aug 28. PMID 31491622
- [Background] Taub ES, Hoffman RS, Manini AF. Incidence and risk factors for hyperlactatemia in ED patients with acute metformin overdose. Am J Emerg Med. 2019 Dec;37(12):2205-2208. doi: 10.1016/j.ajem.2019.03.033. Epub 2019 Mar 23. PMID 30967322